CLINICAL TRIAL: NCT00576004
Title: Pelvic Organ Prolapse Repair With or Without Concomitant Burch Colposuspension in Patients With Urinary Incontinence: A Randomised Surgical Trial
Brief Title: Pelvic Organ Prolapse Repair With or Without Concomitant Burch Colposuspension in Patients With Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Of Perugia (Other)
Responsible Party: Department of Medical-Surgical Specialties and Public Health, Section of Urology and Andrology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC_ML_001; EC_ML_001s
Record Dates: First submitted 2007-12-17; First posted 2007-12-18 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2007-12

CONDITIONS: Pelvic Organ Prolapse; Urinary Incontinence
Keywords: Pelvic organ prolapse, Urinary incontinence, Burch colposuspension, surgery
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A (Active Comparator): Pelvic organ prolapse repair plus concomitant Burch Colposuspension
  Interventions: Procedure: Pelvic organ prolapse repair and Burch colposuspension
- group B (Active Comparator): Pelvic organ prolapse without Burch colposuspension
  Interventions: Procedure: Pelvic organ prolapse repair and Burch colposuspension

INTERVENTIONS:
Procedure: Pelvic organ prolapse repair and Burch colposuspension — Abdominal pelvic organ prolapse repair and retropubic Burch colposuspension

SUMMARY:
To evaluate the impact of Burch colposuspension (BC), as an anti-incontinence measure, in patients with urinary incontinence (UI) undergoing abdominal surgery for pelvic organ prolapse (POP) repair

DETAILED DESCRIPTION:
Forty-seven women suffering from POP and UI were randomly assigned to abdominal POP repair and concomitant BC ( 24 patients; group A) or POP repair alone without any anti-incontinence procedure ( 23 patients.; group B). They were followed-up at 3, 6, and 9 months after surgery and then annually. The primary outcome measures were anatomical outcome and changes in incontinence status as indicated by a bladder diary, the number of daily pads and the stress test. Secondary endpoints were changes in subjective symptoms and Quality of Life (QoL) as measured by the Urogenital Distress Inventory (UDI-6) and the Impact Incontinence Quality of Life (IIQ-7) questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Study inclusion criteria were POP > 2, UI as was defined by ICS [2], age ≥ 18 and ≤ 75 yrs.

Exclusion Criteria:

* Benign or malignant uterus lesion (leiomyoma, fibromyoma, cervical or endometrial carcinoma)
* Active pelvic inflammatory disease,
* Known hypersensitivity to synthetic materials (polypropylene, polythetrafloroethilene, polyethileneterephtalate, polyglactil acid or polyglycolic acid)
* Pregnancy or lactation
* Evidence of clinically significant cardiovascular, renal, hepatic or respiratory diseases; and
* Any condition that in the judgment of the investigators would interfere with the subject's ability to provide informed consent, comply with study instructions, place the subject at increased risk, or which might confound interpretation of study results.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2002-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
changes in the incontinence rate as shown by a bladder diary, number of daily pads and the stress test. | 2002-2006

SECONDARY OUTCOMES:
changes in subjective symptoms and Quality of Life (QoL) as measured by questionnaires | 2002-2206

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Costantini, MD, Principal Investigator — University Of Perugia
Locations (1):
- University of Perugia, Perugia, Perugia, Italy

REFERENCES:
- See also: Related Info — http://www.unipg.it